CLINICAL TRIAL: NCT03207828
Title: "Eficacia de la Terapia de activación Conductual Para Pacientes Con Dolor crónico: Ensayo clínico Randomizado"
Brief Title: Testing Interventions for Patients With Fibromyalgia and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Lydia Gomez Perez, Principal Investigator, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FONIS REGULAR 2017_305
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Fibromyalgia; Depression
Keywords: Behavioral activation
MeSH Terms: conditions — Fibromyalgia; Depression

STUDY DESIGN:
Intervention Model Description: Patients with Fibromialgia and mayor depression will be randomized to two treatment conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants: blind to hypothesis and blind regarding which conditions they have been assigned. To mask the condition, participants of both arms will receive the experimental intervention. Control participants will need to wait to receive the intervention. Control participants will know that the time waiting to be attended can vary among participants (and that even participants in the experimental group may have to wait). They also would know that (while waiting to be intervened) participants will need to attend to a series of assessments, and that five month is the longest period they will need to wait. Care providers: blind to all the study aspects but not to its aims. Investigators: blind to the subject treatment assignment and the outcomes. Outcomes assessors: blind to all aspects. Interventionist: blind to hypothesis and outcomes. Research assistant: blind to everything but not to aims and implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral activation group (Experimental): This group will receive usual care for fibromyalgia with comorbid major depression plus in-group behavioral activation.
  Interventions: Behavioral: Behavioral activation; Other: Usual care
- Usual care (Other): This group of participants will only receive usual care for fibromyalgia with comorbid depression.
  Participants will be attended by a Medical Doctor that has a high level of expertise in fibromyalgia (rheumatologist or chronic pain specialist) of the Red Salud Christus, the most important private medical care network in Chile. In this clinic treatment of fibromyalgia includes administering pregabalin and pain killers (avoiding opioids). I addition, muscle relaxant such as cyclobenzaprine can be also administered. In a high proportion of cases (around 42%), antidepressant with analgesic properties, namely duloxetine, is prescribed. In addition, usual care includes derivation to psychiatrist if needed.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Behavioral activation — The Brief Behavioral Activation Treatment for Depression (Lejuez, Hopko, Acierno, Daughters, & Pagoto, 2011; Lejuez, Hopko, LePage, Hopko, and McNeil; 2001) will be used. It aims are (1) to increase engagement with activities associated with pleasure or mastery experiences; (2) decrease engagement with activities that maintain or increase the risk of depression; (3) and remove the barriers that limit the access to gratification. The sessions of therapy are well structured and described in its manual. The protocol was originally designed to be applied individually. However, for the present research, it will be adjusted to be applied in group sessions (5-8 participants). Materials will be also adjusted to be use with Chilean population. Treatment core aspects will not be altered. The treatment will last 10 sessions over two months. Two psychologist trained in behavioral activation will lead the sessions.
  Other Names: Brief behavioral activation for depression
  Arms: Behavioral activation group
Other: Usual care — Participants will be attended by a Medical Doctor that has a high level of expertise in fibromyalgia (rheumatologist or chronic pain specialist) at the Red Salud Christus, the most important private medical care network in Chile. In this clinic the protocol for the treatment of fibromyalgia includes administering pregabalin or gabapentin and pain killer (avoiding opioids). I addition, muscle relaxant such as cyclobenzaprine can be also administered to improve sleep quality. In a high proportion of cases (around 42%), antidepressant with analgesic properties, namely duloxetine, is prescribed. In addition, usual care includes derivation to psychiatrist if needed.

SUMMARY:
Chronic pain is a major health problem. It causes high economic and social costs around the world and severely impairs the quality of life of those who suffer from it. Chronic pain and major depression frequently co-occur. Patients with both conditions have a worse prognosis and higher disability, and their treatment options are scarce. Behavioral activation (BA) may be an especially useful intervention for these patients. This intervention targets mechanisms of action that seem to be common to both disorders. In spite of this, the efficacy of this intervention has not been yet examined in people with both conditions. Therefore, the purpose of the present study is to examine the efficacy of BA compared to usual care among Chilean women with fibromyalgia and mayor depression (N = 90). Women will be randomized to an experimental arm (n = 45) who will receive usual care (UC) for fibromyalgia with comorbid depression plus BA; and a comparison arm, who will receive only UC for fibromyalgia with comorbid depression (n =45). Primary and secondary outcomes will be assessed before, during, and after the intervention, as well as at a three month follow-up. The investigators expect to find that, after treatment, the group receiving BA will experience higher statistical and clinical significant reductions in depressive symptom severity (primary outcome), as well as in their levels of some pain-related variables (namely pain intensity, fibromyalgia impact, pain-related anxiety, catastrophism, and physical health symptoms severity). In addition, the percentage of women in remission from the diagnosis of depression (as well as the percentage of women responding to treatment) will be greater in the experimental arm than in the comparison arm. Also, the percentage of women who show a clinically significant reduction in pain intensity (decreases greater than two units in the pain intensity scale) will be greater in the experimental arm than in the comparison arm. Finally, the investigators hypothesize that the decrease observed in the pain-related variables will be mediated by the decrease observed in depressive symptoms severity. Regarding the outcomes assessed at a three months follow-up, the investigators expect to find that the differences found after treatment between the two arms will be maintained at follow-up. In order to test our hypothesis, Hierarchical Linear Models (HLM) and Cochran-Mantel-Haenszel tests will be performed. The results of these study might contribute to facilitate the integrated treatment of fibromyalgia and depression, and to reduce the burden on the health system due to the lack of effective therapeutic strategies to treat these comorbidity.

DETAILED DESCRIPTION:
Chronic pain is a word-wide major health problem, which seriously affects the quality of life of those who experience it and causes important socio-economical costs (Tsang et al., 2008). According to the results of the last Chilean National Health Survey (2010), 34.2% of Chileans older than 15 years present pain ranging from moderate to severe. The pain experienced by a considerable proportion of these individuals (73.5%) is chronic. Among Chileans, chronic pain has been found to be related to more sickness leaves, a five-time increase in the use of primary care services, and the presence of depressive disorders (Miranda et al., 2013). In fact, around 35% patients with chronic pain suffer from depression (Gracely, Ceko, & Bushnell, 2012). In the case of some specific pain disorders such as fibromyalgia, this comorbidity is even greater (life prevalence around 90% for depressive symptomatology and 62-86% for major depressive disorder; Gracely et al., 2012). As a result, some authors posit that fibromyalgia and depression are two manifestations of a single affective spectrum disorder (Gracely et al., 2012). In fact, according to some evidence, both disorders share pathophysiological aspects. For example, pharmacological treatment of both fibromyalgia and depression includes the same dual serotonergic and noradrenergic agonists, namely, amitriptyline and duloxetine (Maletic & Raison, 2009).

Depressive symptoms impair chronic pain treatment and are associated with a worse chronic pain prognosis (Li, 2015). The increasing and concomitant prevalence of depression and chronic pain represents a burden for the primary care systems. Providing effective and appropriate primary care interventions to address this comorbidity is indeed needed, considering that chronic pain and depression lead to great disability. Taking into account that reducing disability is part of the second strategic objective of the Health Goals of the Decade 2011-2020 for Chile, the design and dissemination of therapeutic strategies aimed at the treatment of these problems is a priority in this country.

Behavioral Activation (BA) is an evidence-based psychological intervention for depression (Cuijpers, Van Straten, & Warmerdam, 2007; Dimidjian, Barrera, Martell, Muñoz, & Lewinsohn, 2011). It has been shown to be as effective as comprehensive cognitive behavioral therapy (Cuijpers et al., 2007) and antidepressant therapy (Dimidjian et al., 2006), with a lower dropout rate than the latter (Dimidjian et al., 2006). There is also evidence that BA works as well as medication and better than cognitive behavioral therapy in the treatment of severe depression (Dimidjian et al., 2006). Moreover, several meta-analyses support the efficacy of BA for the treatment of depression (Cuijpers et al., 2007; Ekers, Webster, Van Straten, Cuijpers, Richards, & Gilbody, 2014; Mazzucchelli, Kane, & Rees, 2009). According to the result of the last meta-analysis conducted (Ekers et al., 2014) - in which 26 randomized controlled trials (RCTs) were analyzed with a total of 1,524 participants - the treatment with BA is superior to the control condition (usual treatment, placebo, or waiting list), showing a high effect size (standardized mean difference, SMD: -0.74, 95% CI -0.91 a - 0.56). In addition, the examination of four RCTs with 283 participants showed that CT is also superior to medication. In this case the effect size was moderate (SMD -0.42, IC -0.83 to -0.00). Finally, according to the results of different studies conducted with several populations, BA can be used in multiple contexts and populations (Dimidjian et al., 2011) such as adolescents (Jacob, Keeley, Ritschel, and Craighead, 2013), seniors (Quijano et al., 2007), university students (Gawrysiak, Nicholas, & Hopko, 2009), and primary care patients (Uebelacker, Weisberg, Haggarty, & Miller, 2009).

More research on the efficacy of BA is still needed, especially with regard to its effect after follow-up; however the results reported so far are promising. Furthermore, BA is much easier to apply and disseminate than other psychological treatments. For these reasons, there is now an increasing interest in examining the efficacy of this intervention in populations with different comorbidities such as obesity, cancer, anxiety, borderline personality, substance abuse, childhood abuse history, smoking, and post-traumatic stress disorder, among others (Dimidjian et al., 2011).

BA could be particularly suitable for treating depression among patients with chronic pain, as some of its main purposes are fighting inactivity, increasing environmental reinforces, and decreasing aversive experiences. Indeed, inactivity, loss of reinforces, and excessive unpleasant experiences seem to play a key role in the etiology of both depressive disorders and chronic pain (Dimidjian et al., 2011, Leeuw et al. 2007). According to Lewinsohn's integrative model of depression (Lewinsohn, Hoberman, Teri, & Hautzinger, 1985), when a person with certain vulnerabilities faces a stressful event, that event and the emotions associated with it interrupt their normal behavior patterns, reduce the availability of the reinforcers in the environment, and increase the rate of aversive experiences. All this finally leads to depression. Depressive symptoms have a series of behavioral, cognitive, and emotional correlates that make the subject more vulnerable to new stressful events, thus creating a pathological cycle that is self-perpetuating in time. Something similar occurs when a person suffers a painful injury. According to Vlayen and Linton's Fear and Avoidance Model (FAM, 2000), in the face of a painful injury, vulnerable individuals (with increased pain catastrophizing or increased pain-related fear) develop strategies aimed at avoiding pain and the activities that cause it. This leads to inactivity, loss of reinforcers, disability, and depression, and consequently, to the exacerbation of the pain intensity and pain-related anxiety and catastrophizing. The patient is trapped in a vicious circle of symptoms that feed-back each other and perpetuate over time. Taking into account the FAM assumptions, as well as the purpose of the BA, this treatment may likely not only be useful for reducing depression in patients suffering from pain, but also for reducing the intensity of their pain and the anxiety and catastrophism associated with it. BA could break the chain of perpetuation in both disorders. In fact, there are preliminary data that support this premise. In a case study, in which BA was used with a woman who had been suffering from chronic pain associated with a diagnosis of fibromyalgia for 11 years, a clinically significant decrease in depressive symptoms was observed after treatment. In addition, the degree in which the pain interfered with the patient's daily activities was reduced (in a 100%), as well as pain-related anxiety and the use of pain medication use. These results (with the exception of reduction in medication use) were maintained within three months of the intervention (Lundervold, Talley, & Buermann, 2006). These same authors replicated these findings in another study, in which they applied the same treatment to another woman who had been suffering from fibromyalgia for 22 years. In this case, the decreases of pain intensity, pain-related anxiety, depression, and medication use were maintained three and six months after the intervention (Lundervold, Talley, & Buermann, 2008).

Behavioral activation is part of some cognitive behavioral pain management treatments (Ehde, Dillworth, & Turner, 2014) that include - in addition to BA - cognitive re-structuring. There is evidence that such treatments are effective in reducing symptoms associated with chronic pain (Ehde et al, 2014; Williams, Eccleston, & Morley, 2012). The size of the effect of such treatments varies from small to moderate, depending on the outcome variable analyzed. Thus, according to the results of the meta-analysis conducted by Williams and colleagues (2012), compared with the usual treatment, cognitive-behavioral interventions developed for pain management have small but significant effects on pain (SMD = -0.21, CI 95% CI = -0.37 to -0.05, Z = 2.35, p <0.05) and disability (DME = - 0.26, CI 95% = -0.47 a -0.04, Z = 2.35, p < 0.05), and moderate effects on mood (DME = -0.38, 95% CI = -0.57 to -0.18, Z = 3.84, p <0.01) and catastrophism (DME = -0.53, 95% CI = -0.76 to -0.31, Z = 4.58, P <0.01). However, in relation to other active treatments, their effects on disability (DME = -0.19, 95% CI = -0.33 to -0.05, Z = 2.66, p <0.01) and catastrophism (SMD = -0.18, 95 % = -0.36 to 0.00, Z = 1.92, p = 0.05) appear to be small, and no significant effects have been found for pain and mood. In addition, further studies are needed to examine the active components of cognitive behavioral therapy for pain (Ehde et al., 2014). Although BA may be one of the effective components of cognitive behavioral therapy, the intensity and emphasis placed on behavioral activation within cognitive behavioral treatments is small, and is generally limited to use in one session, so it is not known yet whether BA in isolation could have beneficial effects on pain. Furthermore, to our knowledge, no studies have been conducted to examine the efficacy of BA to reduce depressive symptoms in patients with chronic pain (beyond the abovementioned case studies).

Finally, it is important to highlight that BA has multiple advantages that make it very efficient in terms of costs and benefits. First, it is a brief therapy, very easy to apply and disseminate (Dimidjian et al., 2011). In addition, it can be implemented by non-psychologists after appropriate training (e. g., nurses or social workers; Ekers, Richards, McMillan, Bland, & Gilbody, 2011). It can also be implemented in group format (Houghton, Curran, & Saxon, 2008; Porter, Spates, & Smitham, 2004) and in the context of primary care (Dimidjian et al., 2011). Finally, there are preliminary results that support its effectiveness in the Latino population (Bianchi & Henao, 2015; Kanter, Santiago-Rivera, Rusch, Busch, & West, 2010). Taken together, these advantages make BA of particular interest in the Latin American context, where economic limitations often do not allow for long and complex treatments, and access to trained therapists is usually limited. Therefore, the purpose of the present study is to examine the effectiveness of BA in a sample of Chilean women with chronic pain and comorbid mayor depression. For several reasons, the investigators will study the efficacy of this treatment in women with the same diagnosis of chronic pain, namely fibromyalgia. First, because this is the first RCT examining the efficacy of BA in patients with chronic pain, it is advisable to include patients with the same diagnosis to increase the homogeneity of the sample. Secondly, BA may be more effective in this type of patients, as there is a high comorbidity between fibromyalgia and depression and both disorders have been hypothesized to be manifestations of a single affective spectrum disorder (Gracely et al., 2012), Finally, preliminary results on the effects of BA in patients with pain have been reported in women with fibromyalgia.

The investigators expect to find that, after treatment, the women in the experimental arm will experience greater decreases in depressive symptoms severity as well as in the pain-related variables assessed (pain intensity, fibromyalgia impact, pain-related anxiety, catastrophism, and physical health symptoms severity) than women in the comparison arm. In addition, the percentage of women in remission from the diagnosis of depression (as well as the percentage of women responding to treatment) will be greater in the experimental arm than in the comparison arm. Similarly, the percentage of women who show a clinically significant reduction in pain intensity (decreases greater than two units in the pain intensity scale) will be greater in the experimental arm than in the comparison arm. Finally, the investigators hypothesize that the decreases observed in the pain-related variables will be mediated by decreases observed in depressive symptoms severity.

Regarding the outcomes assessed at a three months follow-up, the investigators expect to find that the differences found between the two groups in the depressive symptoms severity and the pain-related variables decreases will be maintained at follow-up. Furthermore, at follow-up the percentage of women in remission from the diagnosis of depression (as well as the percentage of women responding to treatment) will continue to be greater in the experimental arm than in the comparison arm. Similarly, after follow-up, the percentage of women who show a clinically significant reduction in pain intensity will continue to be greater in the experimental arm than in the comparison arm. The differences found after the follow-up in the pain-related variables will be mediated by the differences found in depressive symptoms severity.

Method

Participants:

Women diagnosed with fibromyalgia and major depression attended at the Service of Family Medicine, Reumathology or Traumatology of the UC-Christus Health Network (N = 90) will participate.

The study sample size was calculated for a Hierarchical Linear Model (HLM) in which the primary outcome (changes in depressive symptoms severity) was the dependent variable. Using Mplus, the investigators determined that a sample of 90 participants was needed to reach a power of .80. In this power analysis, the correlation between the intercept and the slope was specified to be -0.4. The average slope was assumed to be negative, as depression scores are expected to drop, and was specified as -0.5. To simplify the model, the variances of the intercept, slope, and scores of all the variables in the model (depressive symptoms severity, and covariates) were specified as 1, so as to have the standardized model solution. The treatment effect on the slope (standardized Beta) was specified as 0.45. This corresponds to a medium-to-large effect size (Cohen, 1992). In addition, the effect of two covariates was included. The effect of each of the covariates on the slope was specified as 0.1. The correlation between treatment and each covariate was specified as 0.1, and the correlation between covariates was specified as 0.3.

Design The present study is a randomized clinical trial with a parallel design. After the diagnosis interview, participants will be randomly assigned to two intervention arms: an experimental arm - that will be treated with BA in a group setting in addition to usual care (UC) for fibromyalgia and comorbid depression- and a comparison arm that will receive only UC for fibromyalgia with comorbid depression. The research design is longitudinal and mixed (within and between subjects repeated measures). Outcomes will be assessed in both groups before, during and after the intervention, as well as after a three-month follow-up, by a research assistant who will be blind to group assignment.

Procedure Participants will be recruited through several procedures. First, posters and brochures with information about the study will be available at the medical attention boxes, so that patients interested in participation could contact the research team by email or phone. In addition, one of the nurses of the medical center will contact by phone all the fibromyalgia patients registered in the medical center to ask them for permission to put them in contact with the study research team. Participants who agree to be contacted will received a phone call by a research assistant, who will provide them with further information about the study and - in order to corroborate that they indeed meet the inclusion criteria for fibromyalgia and mayor depression -ask them to respond to the Fibromyalgia Survey Questionnaire (FSQ; Wolfe et al., 2011; Carrillo de la Peña et al., 2015) and the Patients Health Questionnaire-9 (PHQ-9; Baader et al., 2008). Participants who meet inclusion criteria will be scheduled for a diagnoses interview according to Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria. The Mini-International Neuropsychiatric Interview (MINI; Ferrando, Bobes, & Gilbert, 1999; Sheehan & Lecrubier, 1999) will be applied in order to make the diagnoses. In addition, the Mini-Mental State Examination (Folstein, Folstein, & Mchugh, 1975, González-Hernández et al., 2009) will be administered. All participant will be asked for informed consent before participation. Participants who meet all the inclusion criteria after this interview will be randomized to the two arms. Randomization will be conducted by a research assistant (other than those who will perform the assessments, treatment and data analysis) using a computer program. As a compensation, patients will receive gift card (with a value of 10.000 Chilean pesos) after each outcome assessment interview.

Data analyses In order to test whether there are differences between the groups in the sociodemographic and clinical characteristics assessed at baseline, Student's t-tests will be performed for continuous variables and Chi-square test for categorical variables. If there are small or empty cells in the categorical tests, the Chi-square test will be replaced by an Exact Fisher's Test. Those variables in which statistically significant differences are found will be introduced in the analyses as covariates.

In order to examine the differences between the groups in the reduction of the primary and secondary outcome, HLM will be performed using MPlus. This analysis involves two levels of analysis: intra-subject (Level 1, which analyzes the change of subjects over time) and inter-subject (Level 2, through which the effect of treatment is examined). Repeated measures of symptoms are nested in each subject, and the analysis allows estimating a change parameter along repeated measurements. The analysis tests whether the change parameter varies according to the treatment group, and other covariates. HLM allows to consider in the analyses all participants (including those who abandoned the study). Therefore, these analyses will be conducted according to the principle of intention to treat.

In order to examine whether there are differences between the groups in the remission of the diagnosis of depression, the investigators will perform two Cochran-Mantel-Haenszel tests (one for the results obtained after the intervention and another for the results obtained after the follow-up). Similarly, in order to examine whether there is a response to treatment (reduction of at least 50% in the severity of depressive symptoms; Dimidjian et al., 2006), two other Cochran-Mantel-Haenszel testse will be carried out. Finally, in order to examine whether there are any differences between the groups in the percentage of women responding to treatment with regard to the intensity of pain, two more Cochran-Mantel-Haenszel tests will be performed. Treatment response will be considered if there are reductions of at least two units on the pain scale from 0 to 10, as this is the criteria usually employed for clinically significant pain improvement (Michener, Snyder, & Leggin, 2011). Finally, in order to test whether the decreases found after the follow-up in the pain-related variables are mediated by the decrease in depressive symptoms severity, regression analysis with bootstrapping will be conducted (Preacher & Hayes, 2008).

ELIGIBILITY:
Inclusion criteria:

1. Being 18 years old or older
2. Understanding Spanish
3. Meeting the diagnostic criteria for fibromyalgia according to the Fibromyalgia Survey Questionnaire (FSQ)
4. Have a primary diagnosis of major depression according to the MINI International Neuropsychiatric Interview (MINI).
5. Being receiving usual care for fibromyalgia and depression in the Medical Center San Joaquín (Red Salud UC Christus, Santiago Chile).
6. Being under treatment with duloxetine.

Exclusion criteria:

1. Having past or present history of psychosis, bipolar disorder, or substance use disorder
2. Presenting risk of suicide according to the suicide module of the MINI
3. Presenting a lower score than the cut-off point in the Minimental Cognitive Examination
4. Being participating simultaneously in another therapy for the depression or pain
5. Being treated with antidepressants other than duloxetine
6. Being diagnosed with Rheumatoid arthritis or other connective tissue diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-09-09 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms severity | Depressive symptoms will be assessed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up. As such the participant will be assessed during five months.
  Patients Health Questionnaire-9 (PHQ-9; Baader et al., 2008). It consists of 9 items evaluating the presence of depressive symptoms in the last two weeks. Its psychometric properties have been examined in Chilean population. It shows a sensitivity of 92% and specificity of 89%. Item response options are: 0 = never, 1 = some days, 2 = more than half the days and 3 = almost every day. Patients can be classified in:
  Major depressive syndrome: presence of 5 or more of the 9 depressive symptoms with an index of severity of more than half of the days, and one of the symptoms is mood depressive or anhedonia.
  Other depressive syndrome: presence of 2, 3 or 4 depressive symptoms for more of half the days and one of the symptoms is depressive mood or anhedonia.
  Positive depressive symptoms: presence of at least one or two of the symptoms depressive, but fails to complete the above criteria.
  Negative depressive symptoms: does not present any diagnostic criteria more than half of the days.

SECONDARY OUTCOMES:
Changes in pain intensity | Pain intensity will be assessed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up. As such the participant will be assessed during five months.
  The Composed Pain Intensity Index (Jensen, Turner, Romano, & Fisher, 1999) will be used to assess pain intensity. According to the recommendations of Jensen et al. (1999), patients will be asked to rate their lowest, medium, and strongest pain during the previous week, as well as their current pain, on a scale ranging from 0 (not at all) to 10 (extremely painful). The mean of these four scores will be calculated to obtain the average pain intensity. These scale have shown to be valid and reliable and to be sensible to treatment effects in several studies (Williamson & Hoggart, 2005).
Changes in physical functioning and fibromyalgia symptoms severity. | The FIQ-R will be completed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up.
  The Fibromyalgia Impact Questionnaire Revised (FIQ-R; Bennett et al., 2009) will be used. It comprises 21 items with responses options ranging from 0 to 10, which are organized in three subscales: The functioning scale (9 items), the symptoms scale (10 items), and the general impact subscale (2 items). The functioning scale assess difficulties to performed several activities during last week. The symptoms scale includes items assessing the severity of ten symptoms that frequently affect patients with fibromyalgia (e. g., memory problems, body stiffness, etc). Finally, two items assesses the general impact of the fibromyalgia.
Changes in pain catastrophizing | The PCS will be completed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up.
  Pain Catastrophizing Scale (PCS; Sullivan, Bishop, & Pivik; 1995; García-Campayo, Rodero, Alda, Sobradiel, Montero, et al., 2008). The PCS is one of the most frequently employed scales to assess pain catastrophizing. It comprises 13 items regarding catastrophic pain-related thoughts and emotions that are organized in three subscales: rumination, magnification, and helplessness. Each item has five response options going from 0 Nothing to 4 All the time. The validity and reliability of the PCS has been boadly described in clinical and not clinical samples. The Spanish Scale has properties similar to the original one (García-Campayo et al., 2008).
Changes in pain hypervigilance. | The PVAQ will be completed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up.
  The Spanish version of the Pain Vigilance and Awareness Questionnaire (PVAQ, Esteve et al., 2014) will be used to assess pain related anxiety, specifically its cognitive aspects (namely pain hypervigilance). It comprises nine items organized in two subscales: Active vigilance and active awareness. This questionnaire excellent internal consistency (Cronbach alpha values between .82 and .92) and has proved to be valid.
Changes in self-reported physical health symptoms. | The PHQ-15 will be completed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up.
  Patients Health Questionnaire (PHQ-15; Ros-Moltalbán, Comas-Vives, & García-García, 2010) will be used to assess physical health symptoms. It comprises 15 items inquiring about somatic symptoms, which account for more than 90% of the symptoms reported in outpatient settings. Respondents rate the severity of each symptom on a 3-point scale (i.e., 0=Not bothered at all, 1=Bothered a little, 2 = Bothered a lot). The PHQ-15 enables classification of participants into four categories according to the reported severity of their symptoms: minimal (scores = 0-4), low (scores = 5-9), medium (scores = 10-14), and high (scores = 15-30). The PHQ-15 has excellent internal reliability and adequate convergent validity. It has shown to be useful to assess somatic complains in speaking Spanish sample.
Changes in environmental reward | The RPI will be completed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up.
  The Reward Probability Index, RPI (Carvalho, Gawrysiak, Hellmuth, McNulty, Magidson, Lejuez & Hopko, 2011). It comprises 20 ítems which assess access to environmental reward and are organized in two factors: Reward Probability and Environmental Suppressors) with strong internal consistency (α=.90). The instruments have shown adequate convergent and discriminant validity (Carvalho et al., 2011).

OTHER OUTCOMES:
Changes in pain interference | Pain interference will be assessed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up
  Pain interference will be assessed with the Pain Interference scale of the Spanish version of the Brief Pain Inventory (Ares et al., 2014). This scale comprises seven items each assessing level of interference with function caused by pain in a specific area of life (general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life) in a rating scale going from 0 (no interference) to 10 (complete interference). This scale has shown to present adequate psychometric properties.
Changes in activation | Activation will be assessed four times: at baseline, during treatment (one month after the start of the treatment), immediately after the treatment, and at three month follow up
  Activation will be assessed with the Activation subscale of the Behavioral Activation for Depression Scale (BADS, Barraca, Pérez-Álvarez, & Bleda, 2011). The BADS (Kanter, Mulick, Busch, Berlin, & Martell, 2007) is an instrument aimed at measure changes in avoidance and activation over the course of the BA therapy. In a recent study conducted with Latino participants with depression, a behavioral activation intervention was found to produce higher decreases in depressive symptoms than supporting counselling, but also increased activation and environmental reward (Collado, Calderón, MacPherson, & Lejuez, 2017). The Cronbach alpha for the Activation subscale is .81.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gómez Pérez, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Red Salud UC Christus, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Andres Ares J, Cruces Prado LM, Canos Verdecho MA, Penide Villanueva L, Del Valle Hoyos M, Herdman M, Traseira Lugilde S, Velazquez Rivera I. Validation of the Short Form of the Brief Pain Inventory (BPI-SF) in Spanish Patients with Non-Cancer-Related Pain. Pain Pract. 2015 Sep;15(7):643-53. doi: 10.1111/papr.12219. Epub 2014 Apr 28. PMID 24766769
- [Background] Baader T, Molina JL, Venezian S, Rojas C, Farías R, Fierro-Freixenet C,.. & Mundt C. Validación y utilidad de la encuesta PHQ-9 (Patient Health Questionnaire) en el diagnóstico de depresión en pacientes usuarios de atención primaria en Chile. Rev Chil Neuro-psiquiatr [internet], 2012 Mar [cited 2017 Jul 5]; 50(1): 10-22. Avaliable from: http://www.scielo.cl/scielo.php?pid=S0717-92272012000100002&script=sci_arttext
- [Background] Barraca J, Perez-Alvarez M, Lozano Bleda JH. Avoidance and activation as keys to depression: adaptation of the Behavioral Activation for Depression Scale in a Spanish sample. Span J Psychol. 2011 Nov;14(2):998-1009. doi: 10.5209/rev_sjop.2011.v14.n2.45. PMID 22059343
- [Background] Costa C, Pinto AM, Pereira AT, Marques M, Macedo A, Pereira da Silva JA. Psychometric properties of the Revised Fibromyalgia Impact Questionnaire (FIQR) - a contribution to the Portuguese validation of the scale. Acta Reumatol Port. 2016 Jul-Sep;41(3):240-250. PMID 27683063
- [Background] Bianchi J, Henao A. Activación conductual y depresión: Conceptualización, evidencia y aplicaciones en Iberoamérica. Ter Psicolo [internet] 2015 May 12 [cited 2017 Jul 5]; 33(2): 69-80. Available from: http://www.scielo.cl/pdf/terpsicol/v33n2/art02.pdf
- [Background] Carrillo-de-la-Pena MT, Trinanes Y, Gonzalez-Villar A, Romero-Yuste S, Gomez-Perretta C, Arias M, Wolfe F. Convergence between the 1990 and 2010 ACR diagnostic criteria and validation of the Spanish version of the Fibromyalgia Survey Questionnaire (FSQ). Rheumatol Int. 2015 Jan;35(1):141-51. doi: 10.1007/s00296-014-3074-3. Epub 2014 Jun 22. PMID 24952419
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Collado A, Castillo SD, Maero F, Lejuez CW, Macpherson L. Pilot of the brief behavioral activation treatment for depression in latinos with limited english proficiency: preliminary evaluation of efficacy and acceptability. Behav Ther. 2014 Jan;45(1):102-15. doi: 10.1016/j.beth.2013.10.001. Epub 2013 Oct 16. PMID 24411118
- [Background] Cuijpers P, van Straten A, Warmerdam L. Behavioral activation treatments of depression: a meta-analysis. Clin Psychol Rev. 2007 Apr;27(3):318-26. doi: 10.1016/j.cpr.2006.11.001. Epub 2006 Dec 19. PMID 17184887
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Dimidjian S, Barrera M Jr, Martell C, Munoz RF, Lewinsohn PM. The origins and current status of behavioral activation treatments for depression. Annu Rev Clin Psychol. 2011;7:1-38. doi: 10.1146/annurev-clinpsy-032210-104535. PMID 21275642
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Ehde DM, Dillworth TM, Turner JA. Cognitive-behavioral therapy for individuals with chronic pain: efficacy, innovations, and directions for research. Am Psychol. 2014 Feb-Mar;69(2):153-66. doi: 10.1037/a0035747. PMID 24547801
- [Background] Ekers D, Richards D, McMillan D, Bland JM, Gilbody S. Behavioural activation delivered by the non-specialist: phase II randomised controlled trial. Br J Psychiatry. 2011 Jan;198(1):66-72. doi: 10.1192/bjp.bp.110.079111. PMID 21200079
- [Background] Ekers D, Webster L, Van Straten A, Cuijpers P, Richards D, Gilbody S. Behavioural activation for depression; an update of meta-analysis of effectiveness and sub group analysis. PLoS One. 2014 Jun 17;9(6):e100100. doi: 10.1371/journal.pone.0100100. eCollection 2014. PMID 24936656
- [Background] Esteve R, Ramirez-Maestre C, Lopez-Martinez AE. Empirical evidence of the validity of the Spanish version of the pain vigilance awareness questionnaire. Int J Behav Med. 2013 Mar;20(1):59-68. doi: 10.1007/s12529-011-9216-z. PMID 22205550
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gawrysiak M, Nicholas C, Hopko DR. Behavioral activation for moderately depressed university students: Randomized controlled trial. J Couns Psychol [internet]. 2009 Jul; 56(3): 468. Available From: http://dx.doi.org/10.1037/a0016383
- [Background] González-Hernández J, Aguilar L, Oporto S, Araneda L, Vásquez M, Von Bernhardi R. Normalización del "Mini-Mental State Examination" según edad y educación, para la población de Santiago de Chile. Rev. Memoriza [internet] 2009 [cited 2017 Jul 5]; 3:23-34. Available From: http://www.memoriza.com/documentos/revista/2009/minimental2009_3_23-34.pdf
- [Background] Gracely RH, Ceko M, Bushnell MC. Fibromyalgia and depression. Pain Res Treat. 2012;2012:486590. doi: 10.1155/2012/486590. Epub 2011 Nov 19. PMID 22191023
- [Background] Houghton S, Curran J, Saxon D. An uncontrolled evaluation of group behavioral activation for depression. Behavior and Cog Psych [Internet] 2008 Mar [cited 2017 Jul 5]; 36: 235-39. Available from: https://www.cambridge.org/core/services/aop-cambridge-core/content/view/CF303D2B68B4E01C8BB90BC216073C3B/S1352465808004207a.pdf/an_uncontrolled_evaluation_of_group_behavioural_activation_for_depression.pdf
- [Background] Jacob M, Keeley ML, Ritschel L, Craighead WE. Behavioural activation for the treatment of low-income, African American adolescents with major depressive disorder: a case series. Clin Psychol Psychother. 2013 Jan-Feb;20(1):87-96. doi: 10.1002/cpp.774. Epub 2011 Aug 22. PMID 21861272
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Leeuw M, Goossens ME, Linton SJ, Crombez G, Boersma K, Vlaeyen JW. The fear-avoidance model of musculoskeletal pain: current state of scientific evidence. J Behav Med. 2007 Feb;30(1):77-94. doi: 10.1007/s10865-006-9085-0. Epub 2006 Dec 20. PMID 17180640
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Hopko DR, Lejuez CW, LePage JP, Hopko SD, McNeil DW. A brief behavioral activation treatment for depression. A randomized pilot trial within an inpatient psychiatric hospital. Behav Modif. 2003 Sep;27(4):458-69. doi: 10.1177/0145445503255489. PMID 12971122
- [Background] Lewinsohn PM, Hoberman H, Teri L, Hautzinger M. An integrative theory of depression. In Theoretical Issues in Behavior Therapy, Ed. S. Reiss, R. Bootzin, pp. 331-59. New York: Academic, 1985. http://www.cambridge.org/cl/academic/subjects/medicine/mental-health-psychiatry-and-clinical-psychology/cambridge-textbook-effective-treatments-psychiatry?format=HB&isbn=9780521842280#jXZHiZM5XTIExWXK.97
- [Background] Li JX. Pain and depression comorbidity: a preclinical perspective. Behav Brain Res. 2015 Jan 1;276:92-8. doi: 10.1016/j.bbr.2014.04.042. Epub 2014 May 2. PMID 24797835
- [Background] Lundervold DA, Talley C, Buermann M. Effect of Behavioral Activation Treatment on fibromyalgia-related pain anxiety cognition. Int J Behav Consult Ther [Internet] 2006 [cited 2017 Jul 5]; 2(1):73, 2006. Available from: http://psycnet.apa.org/journals/bct/2/1/73.pdf
- [Background] Lundervold DA, Talley C, Buermann M. Effect of behavioral activation treatment on chronic fibromyalgia pain: Replication and extension. Int J Behav Consult Ther [Internet] 2008 [cited 2017 Jul 5]; 4(2):146 - 157. Available from: http://psycnet.apa.org/journals/bct/4/2/146.pdf
- [Background] Encuesta Nacional de Salud Chile. ENS 2009-2010. Tomo V: Resultados. Available from: http://web.minsal.cl/portal/url/item/bcb03d7bc28b64dfe040010165012d23.pdf
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827
- [Background] Ferrando L, Bobes J, Gilbert J, Soto, M, Soto, O. Mini International Neuropychiatric Interview (M.I.N.I.). Versión en Español 5.0.0. Madrid: Instituto IAP, 2000. Available from: http://www.academia.cat/files/425-7297-DOCUMENT/MinientrevistaNeuropsiquatribaInternacional.pdf
- [Background] Kanter JW, Santiago-Rivera AL, Rusch LC, Busch AM, West P. Initial outcomes of a culturally adapted behavioral activation for Latinas diagnosed with depression at a community clinic. Behav Modif. 2010 Mar;34(2):120-44. doi: 10.1177/0145445509359682. Epub 2010 Feb 22. PMID 20176914
- [Background] Mazzucchelli T, Kane R, Rees C. Behavioral activation treatments for depression in adults: a meta-analysis and review. Clin Psych: Science Prac [Internet] 2009 [cited 2017 Jul 05]; 16(4):383-411. Available from: http://onlinelibrary.wiley.com/doi/10.1111/j.1468-2850.2009.01178.x/epdf
- [Background] Miranda JP, Quezada P, Caballero P, Jiménez L, Morales A, Bilbeny N, Vega JC. Revisión Sistemática: Epidemiología de Dolor Crónico No Oncológico en Chile. Rev El Dolor [Internet] 2013 [cited 2017 Jul 05]; 59: 10-17. Available from: http://www.ached.cl/upfiles/revistas/documentos/53dfbe675a347_original1_59.pdf
- [Background] Porter JF, Spates CR, Smitham S. Behavioral Activation Group Therapy in Public Mental Health Settings: A Pilot Investigation. Prof Psychol Res Pr [Internet] 2014 [cited 2017 Jul 05]; 35(3): 297 -301. Available from: http://dx.doi.org/10.1037/0735-7028.35.3.297
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Quijano LM, Stanley MA, Peterson, NJ, Casado BL, Steinberg EH, Cully, JA, Wilson NL. Healthy Ideas: a depression intervention delivered by community-based case managers serving older adults. J Appl Gerontol [Internet] 2007 [cited 2017 Jul 05];26: 139-56. Available from: journals.sagepub.com/doi/pdf/10.1177/0733464807299354
- [Background] Maletic V, Raison CL. Neurobiology of depression, fibromyalgia and neuropathic pain. Front Biosci (Landmark Ed). 2009 Jun 1;14(14):5291-338. doi: 10.2741/3598. PMID 19482616
- [Background] Ros Montalban S, Comas Vives A, Garcia-Garcia M. Validation of the Spanish version of the PHQ-15 questionnaire for the evaluation of physical symptoms in patients with depression and/or anxiety disorders: DEPRE-SOMA study. Actas Esp Psiquiatr. 2010 Nov-Dec;38(6):345-57. Epub 2010 Nov 1. PMID 21188674
- [Background] Sullivan M, Bishop S, Pivik J. The Pain Catastrophizing Scale: Development and Validation. Psychol Assessment [Internet] 1995 [cited 2017 Jul 05]; 7(4): 524-532. Available from: http://dx.doi.org/10.1037/1040-3590.7.4.524
- [Background] Tsang A, Von Korff M, Lee S, Alonso J, Karam E, Angermeyer MC, Borges GL, Bromet EJ, Demytteneare K, de Girolamo G, de Graaf R, Gureje O, Lepine JP, Haro JM, Levinson D, Oakley Browne MA, Posada-Villa J, Seedat S, Watanabe M. Common chronic pain conditions in developed and developing countries: gender and age differences and comorbidity with depression-anxiety disorders. J Pain. 2008 Oct;9(10):883-91. doi: 10.1016/j.jpain.2008.05.005. Epub 2008 Jul 7. PMID 18602869
- [Background] Uebelacker LA, Weisberg RB, Haggarty R, Miller IW. Adapted behavior therapy for persistently depressed primary care patients: an open trial. Behav Modif. 2009 May;33(3):374-95. doi: 10.1177/0145445509331924. Epub 2009 Mar 11. PMID 19282506
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance and its consequences in chronic musculoskeletal pain: a state of the art. Pain. 2000 Apr;85(3):317-332. doi: 10.1016/S0304-3959(99)00242-0. PMID 10781906
- [Background] Williams AC, Eccleston C, Morley S. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD007407. doi: 10.1002/14651858.CD007407.pub3. PMID 23152245
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Background] Carvalho JP, Gawrysiak MJ, Hellmuth JC, McNulty JK, Magidson JF, Lejuez CW, Hopko DR. The reward probability index: design and validation of a scale measuring access to environmental reward. Behav Ther. 2011 Jun;42(2):249-62. doi: 10.1016/j.beth.2010.05.004. Epub 2011 Jan 18. PMID 21496510
- [Derived] Gomez-Perez L, Verges A, Vazquez-Taboada AR, Duran J, Gonzalez Tugas M. The efficacy of adding group behavioral activation to usual care in patients with fibromyalgia and major depression: design and protocol for a randomized clinical trial. Trials. 2018 Nov 29;19(1):660. doi: 10.1186/s13063-018-3037-1. PMID 30486843